CLINICAL TRIAL: NCT06982716
Title: Evaluating the Clinical Effectiveness of a Community-based Hearing Aid Fitting Service Delivery Model Facilitated by Community Healthcare Workers (CHWs) Providing Smartphone-based In-situ and Pre-set Hearing Aid Fittings in Low- and Middle-income Communities (LMICs)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pretoria (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, De Wet Swanepoel, Professor De Wet Swanepoel, University of Pretoria
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4R33DC019598-03 (NIH); 4R33DC019598-03 (NIH)
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss
Keywords: hearing loss; community-based; hearing aid; service delivery model; Community healthcare workers; in-situ; pre-set hearing aids; randomized controlled trial; low- and middle-income
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: A randomized, three-arm, single-blind placebo trial with 90 participants will be used. Randomization will be conducted before participant enrolment ensuring that each participant is assigned to one of the three study arms (In-situ fitting, Pre-set fitting, or Minimal Gain fitting) before enrolling in the study.
  After baseline assessments to determine candidacy (T0), participants will be randomly assigned and start with one of the three interventions (T1). There will be one placebo-control group with Lexie Lumen hearing aids fitted to minimal gain (i.e., 10 dB HL across the frequency range regardless of hearing loss levels) with two experimental groups: (i) In-situ hearing aid fitting using a proprietary algorithm on Lexie Lumen hearing aids that are based on the National Acoustics Laboratories Non-Linear Version 2 (NAL-NL2) algorithm (ii) Pre-set hearing aid fitting with Go Ultra hearing aids. The minimal gain group (control) will be crossed over to the in-situ fitting after 6 weeks
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- In-situ Group (Experimental): * The CHW will fit each participant in the in-situ group with the Lumens programmed using the smartphone-based in-situ (proprietary algorithm based on the NAL-NL2) fitting.
  * Participants will select the listening environment they feel most comfortable with.
  Interventions: Device: Lexie Lumen Hearing Aids
- Control Group (Other): * Participants in the control group will be fitted with Lumens programmed using minimal gain (10 dB gain across frequencies regardless of degree of HL). This will be conducted by the CHW.
  * Participants will select the listening environment they feel most comfortable with.
  Interventions: Device: Lexie Lumen Hearing Aids
- Pre-set Group (Experimental): ● The CHW will fit each participant in the pre-set group with Go Ultra hearing aids on one of the four pre-set programs. Participants will select the program they feel most comfortable with.
  Interventions: Device: Go Ultra Hearing Aids

INTERVENTIONS:
Device: Lexie Lumen Hearing Aids — The Lexie Lumens (Lexie Hearing) are self-fitting wireless air conduction hearing aids consisting of 16 channels, wide-dynamic-range compression technology, feedback reduction, Bluetooth connectivity and programming, digital noise reduction, and a directional microphone array. These hearing aids will be sourced at a cost of $240 USD per pair as this study will be conducted in low-income settings. The hearing aids allow for Bluetooth in-situ hearing aid fitting using the Lexie proprietary fitting algorithm that is based on the NAL/NL2 algorithm from a smartphone application (Lexie Hearing) based on the four hearing thresholds tested. These digital hearing aids were designed for use by adults over the age of 18 years with known or self-perceived mild-to-moderate hearing loss. The Lexie Lumens are behind-the-ear (BTE) hearing aids powered by replaceable batteries. Individuals can conduct an in-situ hearing test via the hearing aids for customized amplification or select a minimal gain.
  Arms: Control Group; In-situ Group
Device: Go Ultra Hearing Aids — Go Ultras (GoHearing) are rechargeable, BTE pre-set hearing aids with advanced audio features, digital sound processing and Bluetooth-streaming capabilities. Designed for adults with mild-to-moderate hearing loss, these hearing aids have four unique programs that the user can manually change to ensure optimal listening comfort. These devices have both program and volume memory functions, as well as noise and wind noise reduction. Go Ultras will be sourced at a cost of less than $130 USD per pair, as this study will be conducted in low-income settings.
  Arms: Pre-set Group

SUMMARY:
The purpose of this study is to advance hearing care in low- and middle-income countries (LMICs) through the rigorous evaluation and optimization of innovative interventions and technologies. This study encompasses the following key aim:

This study aims to establish the effectiveness of community-based hearing aid fittings facilitated by community healthcare workers (CHWs) using mobile health (mHealth) technologies in low- and middle-income communities (LMICs). The primary goal is to determine the efficacy of CHW-facilitated smartphone-based in-situ hearing aid (HA) fittings (a proprietary fitting based on the NAL-NL2 algorithm) and pre-set HAs fittings compared to minimal amplification through a single-blind randomized controlled trial (RCT). By comparing self-reported benefits between the experimental and control groups, this aim seeks to demonstrate the superiority of the CHW-facilitated smartphone-based and pre-set hearing aid fittings compared to minimal amplification.

DETAILED DESCRIPTION:
This study aims to establish the effectiveness of community-based hearing aid fittings facilitated by community healthcare workers (CHWs) using mobile health (mHealth) technologies in low- and middle-income communities (LMICs). The investigators hypothesize that amplification offered by smartphone-based in-situ hearing aid (HA) fittings and pre-set hearing aid fittings facilitated by CHWs have superior self-reported outcomes compared to minimal amplification.

To test this hypothesis, the investigators will conduct a single-blind randomized controlled trial (RCT) where participants are assigned to either the experimental smartphone-based in-situ hearing aid fitting, pre-set hearing aid fitting, or minimal amplification fitting. A minimal amplification fitting provides only the most basic level of amplification without individualized adjustments. This level of amplification is primarily intended to prevent occlusion effects rather than to offer meaningful hearing benefits. In this study, a flat 10 dB gain will be provided across frequencies regardless of the degree of hearing loss. A placebo-controlled design is essential for assessing the true effectiveness of hearing aid interventions beyond non-specific effects such as participant expectations or the general experience of wearing a device. Comparing experimental conditions to minimal amplification ensures that any observed benefits are attributable to the intervention rather than psychological or external influences.

Outcomes will be measured by self-reported benefits, with control participants offered the smartphone-based in-situ fitting after six weeks. All participants will also receive a paper-based hearing aid acclimatization and support programme on the day of the hearing aid fitting to assist them in hearing aid use and maintenance. The participants will also be provided a contact number for the CHWs to contact if any assistance is needed.

Rationale Given the limited access to hearing care in LMICs due to prohibitive costs and scarcity of trained professionals, this study leverages mHealth solutions and task-shifting to CHWs as a sustainable and scalable approach. Preliminary studies have shown promising results for the components of these interventions, justifying the need for clinical trials to evaluate their effectiveness. By focusing on end-to-end smartphone-based in-situ hearing aid fittings and acclimatization support, this study aims to create an innovative and accessible model of hearing care that could significantly reduce the global burden of hearing loss.

Additionally, understanding the difference in outcomes between meaningful amplification and minimal amplification is crucial for guiding hearing care strategies in LMICs. If substantial benefits are observed in the experimental groups relative to minimal amplification, it strengthens the case for scaling up CHW-facilitated hearing aid provision as a cost-effective solution. Conversely, if minimal amplification yields similar self-reported outcomes, it may suggest that additional interventions (e.g., counseling, expectations management) are necessary for maximizing hearing aid benefits in these settings.

A randomized, three-arm, single-blind placebo trial (full blinding details below) with 90 participants will be used. The estimated timeline for trial completion is approximately 52 weeks post-hearing aid fitting. The clinical trial will be conducted across three sites (Khayelitsha and Drakenstein Districts in the Western Cape Province of South Africa and Atteridgeville District in the Gauteng Province of South Africa).

Randomization will be conducted before participant enrollment, ensuring that each participant is assigned to one of the three study arms (In-situ fitting, Pre-set fitting, or Minimal Gain fitting) before enrolling in the study.

After baseline assessments to determine candidacy (T0), participants will be randomly assigned and start with one of the three interventions (T1). There will be one placebo-control group with Lexie Lumen hearing aids fitted to minimal gain (i.e., 10 dB HL across the frequency range regardless of hearing loss levels) with two experimental groups: (i) In-situ hearing aid fitting using a proprietary algorithm on Lexie Lumen hearing aids that are based on the National Acoustics Laboratories Non-Linear Version 2 (NAL-NL2) algorithm (ii) Pre-set hearing aid fitting with Go Ultra hearing aids. Following fitting (T1), there will be a 6-week field trial, with follow-up visits scheduled at 6 weeks (T2). Following that, the minimal gain group (control) will be crossed over to in-situ fitting (CG-T2;), and another 6-week field trial will be conducted (follow up at CG-T3). Follow-up visits for the In-situ and Pre-set groups will occur again at 12 weeks (T3), 26 weeks (T4), and 52 weeks (T5).

The primary endpoint will be at the six-week follow-up. The primary outcome measure will be the IOI-HA. A difference of ≥3 points in the IOI-HA score is considered clinically significant based on prior research by Apple, representing a meaningful improvement in hearing aid benefit, satisfaction, and quality of life.

The secondary measures will be the RHHI-S, SNI, and EQ-5D-5L. Baseline RHHI-S, SNI, and EQ-5D-5L scores will be compared with scores obtained at subsequent follow-up visits.

Additionally, a questionnaire with Likert scale questions targeting functional use and meaningful life changes will be completed at all follow-up visits.

Procedure - All assessment and fitting procedures will be facilitated by the CHWs T0: Baseline assessment

* Assess participants for candidacy
* Obtain Informed Consent from the participants
* Record demographic information
* Complete the baseline EQ-5D-5L, SNI, and RHHI-S
* Conduct otoscopy
* Conduct audiometric evaluation to ensure that participants meet the pure tone air-conduction thresholds to be included.
* The clinical research audiologists will then establish candidacy by reviewing the otoscopy and PTA results. The eligible participants will be randomly allocated to either the In-situ, Control, or Pre-set group. Randomization will be conducted before participant enrollment, ensuring that each participant is assigned to one of the three study arms (Lexie Lumen with in-situ fitting, Go Ultra with Pre-set fitting, or Minimal Gain) before enrolling in the study. A random number generator will allocate participant numbers to the respective arms. As soon as a participant is enrolled, they will automatically be assigned to one of the three arms based on the predefined randomization process. This approach ensures unbiased group allocation from the outset of the study. This randomization will be done by an additional independent party.

T1: Hearing-aid fitting Once randomized into one of the three groups, participants will be booked for Visit 2 for hearing aid fitting. All participants will undergo otoscopy, and the participants (not the pre-set group) will undergo an in-situ hearing test via the Lumen hearing aids before the hearing aid fitting.

In-situ Group

* The CHW will fit each participant in the in-situ group with the Lumens programmed using the smartphone-based in-situ (proprietary algorithm based on the NAL-NL2) fitting.
* Participants will select the listening environment they feel most comfortable with.

Control Group

* Participants in the control group will be fitted with Lumens programmed using minimal gain (10 dB gain across frequencies regardless of degree of HL). This will be conducted by the CHW.
* Participants will select the listening environment they feel most comfortable with.

Pre-set Group

● The CHW will fit each participant in the pre-set group with Go Ultra hearing aids on one of the four pre-set programs. Participants will select the program they feel most comfortable with.

T2: Follow-up #1 and cross-over for Control Group

* After 6 weeks of hearing aid use, participants from all groups will return for a follow-up assessment.
* The International Outcome Inventory for Hearing Aids (IOI-HA), the Revised Hearing Handicap Inventory - Screening (RHHI-S), EQ-5D-5L, SNI, and a non-standardized questionnaire will be completed by the participants.
* The control group will then be offered the in-situ intervention (proprietary in-situ fitting based on NAL-NL2).
* An administrative assistant will collect outcome measures to avoid CHW bias.

T3: Follow-up #2 (Final follow-up for Control Group)

* After 12 weeks of hearing aid use, all participants will return for a follow-up assessment.
* The International Outcome Inventory for Hearing Aids (IOI-HA), the Revised Hearing Handicap Inventory - Screening (RHHI-S), EQ-5D-5L, SNI, and a non-standardized questionnaire will be completed by the participants.
* An administrative assistant will collect outcome measures to avoid CHW bias.

T4: Follow-up #3

* After 26 weeks of hearing aid use, only participants from the Experimental groups will return for a follow-up assessment.
* The International Outcome Inventory for Hearing Aids (IOI-HA), the Revised Hearing Handicap Inventory - Screening (RHHI-S), EQ-5D-5L, SNI, and a non-standardized questionnaire will be completed by the participants.
* An administrative assistant will collect outcome measures to avoid CHW bias.

T5: Final Review

* After 52 weeks of hearing aid use, only participants from the Experimental groups will return for a follow-up assessment.
* The International Outcome Inventory for Hearing Aids (IOI-HA), the Revised Hearing Handicap Inventory - Screening (RHHI-S), EQ-5D-5L, SNI, and a non-standardized questionnaire will be completed by the participants.
* An administrative assistant will collect outcome measures to avoid CHW bias.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Confirmed mild to severe (20 to < 80 dB PTA in both ears; (World Health Organization, 2021)) hearing loss (determined during baseline assessments)
* Willing/available to commit to at least 6- and 12-week follow-ups

Exclusion Criteria:

* Younger than 18 years
* Hearing loss too severe (≥80 dB HL PTA)
* Normal hearing (<20 dB HL PTA)
* Middle ear pathology such as otitis media; active drainage from the ears.
* Unwilling/unavailable to commit to at least 6- and 12-week follow-ups.
* Unilateral hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
International Inventory for Hearing Aids (IOI-HA) | The primary endpoint will be at the six-week follow-up. However, data will be collected at the 6 week, 12 week, 26 week and 52 week follow-up.
  The IOI-HA is a validated seven-item questionnaire to measure the effectiveness of the hearing aid intervention (Cox and Alexander, 2002). It targets seven domains including, (i) daily use, (ii) benefit, (iii) residual activity limitations, (iii) satisfaction, (iv) residual participation restrictions, (v) impact on others, and (vi) quality of life. Each item is scored on a 5-point Likert scale, with higher scores indicating more favorable outcomes. The five response choices range from the worst (score of 1) to best (score of 5) outcome . The IOI-HA has been translated to the languages most commonly used in these communities namely isiXhosa and Sepedi. The participants will have the option to complete the IOI-HA in either of these languages or in English.

SECONDARY OUTCOMES:
Revised Hearing Handicap Inventory and Screening Tool (RHHI-S) | Baseline, 6, 12, 26 and 52 week follow-up
  The RHHI-S is a validated 10-item questionnaire that is a strong unidimensional, clinically informative measure of self-perceived hearing handicap that can be used by adults of all ages (Cassarly, Matthews, Simpson, & Dubno, 2020). Respondents answer each item using a 3-point Likert scale: yes (4 points), sometimes (2 points), or no (0 points). The total score ranges from 0 to 40, with higher scores indicating greater self-perceived hearing handicap. The RHHI-S has been translated into the languages most commonly used in these communities, namely isiXhosa and Sepedi. The participants will have the option to complete the RHHI-S in either of these languages or in English.
EQ-5D-5L | Baseline, 6, 12, 26 and 52 week follow-up
  The EQ-5D-5L is a standardized instrument used to measure generic health-related quality of life. It consists of two components:
  Descriptive System - This includes five dimensions: Mobility, Self-care, Usual activities, Pain/discomfort and Anxiety/depression. Each dimension is rated on a 5-level Likert scale: 1 = No problems to 5 = Extreme problems / Unable to perform. The combination of responses defines a health state, which can be converted into an index value using a country-specific value set. Index scores typically range from less than 0 (health states worse than death) to 1 (perfect health).
  Visual Analogue Scale - A self-rated health score on a vertical scale from 0 (worst imaginable health) to 100 (best imaginable health). The EQ-5D-5L has been translated into the languages most commonly used in these communities, namely isiXhosa and Northern Sotho (Sepedi). The participants will have the option to complete the EQ-5D-5L in either of these languages or in English.
Berman-Syme Social Network Index (SNI) | The SNI will be completed at Baseline for all participants and then at the 6 week, 12 week, 26 week, and 52 week follow-up for participants who received the intervention
  The Berman-Syme Social Network Index (SNI) evaluates participants' social connectedness based on four domains: (1) marital status, (2) frequency and quantity of contact with friends and relatives, (3) participation in religious meetings, and (4) involvement in community or organizational groups. Following the approach outlined by Loucks et al. (2006), responses are converted into binary scores and then summed to create a composite index ranging from 0 to 4. The total score reflects the degree of social integration, with higher scores indicating greater social connectedness.

CONTACTS AND LOCATIONS:
Overall Officials: Professor De Wet Swanepoel, PhD Audiology, Principal Investigator — University of Pretoria
Locations (3):
- South Africa (3):
  - Atteridgeville Community, Pretoria, Gauteng
  - Khayelitsha Community, Cape Town, Western Cape
  - Paarl Valley, Paarl, Western Cape

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loucks EB, Sullivan LM, D'Agostino RB Sr, Larson MG, Berkman LF, Benjamin EJ. Social networks and inflammatory markers in the Framingham Heart Study. J Biosoc Sci. 2006 Nov;38(6):835-42. doi: 10.1017/S0021932005001203. Epub 2006 Jan 27. PMID 16441967
- [Background] Keidser G, Dillon H, Flax M, Ching T, Brewer S. The NAL-NL2 Prescription Procedure. Audiol Res. 2011 Mar 23;1(1):e24. doi: 10.4081/audiores.2011.e24. eCollection 2011 May 10. No abstract available. PMID 26557309
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Cox RM, Rivera IM. Predictability and reliability of hearing aid benefit measured using the PHAB. J Am Acad Audiol. 1992 Jul;3(4):242-54. PMID 1421456
- [Background] Bisgaard N, Zimmer S, Laureyns M, Groth J. A model for estimating hearing aid coverage world-wide using historical data on hearing aid sales. Int J Audiol. 2022 Oct;61(10):841-849. doi: 10.1080/14992027.2021.1962551. Epub 2021 Aug 24. PMID 34428121
- [Background] Arlinger S, Nordqvist P, Oberg M. International Outcome Inventory for Hearing Aids: Data From a Large Swedish Quality Register Database. Am J Audiol. 2017 Oct 12;26(3S):443-450. doi: 10.1044/2017_AJA-16-0123. PMID 29049627

DOCUMENTS (4):
  • Study Protocol (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT06982716/Prot_002.pdf
  • Statistical Analysis Plan (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT06982716/SAP_003.pdf
  • Informed Consent Form: Baseline Informed Consent (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT06982716/ICF_000.pdf
  • Informed Consent Form: Hearing aid fitting informed consent (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT06982716/ICF_001.pdf